CLINICAL TRIAL: NCT03260868
Title: Evaluation of Virtual Versus Traditional Study Conduct in a 6-month, Multicenter, Randomized, Open-label, Two-parallel Group Pilot Study in Adult Patients With Type 1 Diabetes Mellitus
Brief Title: Evaluation of Virtual Versus Traditional Study Conducted in a Group Pilot Study in Adult Patients With Type 1 Diabetes Mellitus (eStudy)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to "prolonged low participant recruitment"
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC15146; U1111-1188-5647 (Other: UTN)
Record Dates: First submitted 2017-08-14; First posted 2017-08-24 (Actual); Results first posted 2020-01-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; Insulin Lispro; Insulin Aspart; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual (Experimental): Participants included in this virtual trial approach group did not visit the study sites during the study course. All study assessments, including vital signs, weight, laboratory variables, etc., were completed via the Bluetooth devices that instantly transfer the digital data.
  Interventions: Drug: Insulin glargine, 300 units per milliliter (U/mL); Drug: Background therapy: Rapid Acting meal time insulin analogs (Humalog, Novolog or Apidra)
- Traditional (Active Comparator): Participants included in this traditional trial approach group visited the study site, followed the study visit schedules for all study assessments that was performed either in-person or phone visits.
  Interventions: Drug: Insulin glargine, 300 units per milliliter (U/mL); Drug: Background therapy: Rapid Acting meal time insulin analogs (Humalog, Novolog or Apidra)

INTERVENTIONS:
Drug: Insulin glargine, 300 units per milliliter (U/mL) — Self-administered subcutaneous injection using prefilled pen once daily for 24 weeks. Dose titration to achieve fasting self-monitoring of plasma glucose (SMPG) level between 80 and 130 milligram per deciliter (mg/dL).
  Other Names: Toujeo ®
Drug: Background therapy: Rapid Acting meal time insulin analogs (Humalog, Novolog or Apidra) — Subcutaneous injection.

SUMMARY:
Primary Objective:

To evaluate the effect of virtual approach via novel technologies versus traditional study conduct on glycemic control in terms of glycated hemoglobin (HbA1c).

Secondary Objective:

To evaluate the appropriate utilization of virtual approach via novel technologies during the study and to assess the effect of the virtual versus traditional study conduct on multiple outcomes in terms of study methodology and diabetes management.

DETAILED DESCRIPTION:
The study had a maximum study duration of 29 weeks, which consisted of a 3-week screening period (including a possible 1-week delay in first investigational medicinal product [IMP] administration after randomization in virtual group due to shipment of IMP and the virtual devices), a 24-week treatment period, and 1-week post-treatment safety follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Participants with Type 1 diabetes mellitus (T1DM) diagnosed at least one year before the screening visit.
* Participants who were treated with multi-dose insulin using insulin glargine 100 U/mL (eg, Lantus or Basaglar) as basal insulin and rapid acting insulin analogues as bolus insulin.
* Participants with access to or experience with mobile technology (eg, tablet or smart phone).
* eSign the consent on the study web portal.

Exclusion criteria:

* Age less than (<) 18 years at screening (Visit 1 - Step 1).
* Type 2 diabetes mellitus.
* HbA1c <5.4 percent (%) or greater than or equal to (>=) 9.0% measured by the central lab at Visit 1.
* Participants who received <6 months treatment with any basal plus (+) meal-time insulin.
* Use of any basal insulins other than insulin glargine 100 U/mL (eg, Lantus or Basaglar) within 3 months before screening.
* Use of an insulin pump within 6 months before screening.
* Use of meal-time insulin other than rapid-acting insulin analogs (Humalog, Novolog, or Apidra), eg, human regular insulin, within 30 days before screening.
* Hemoglobinopathy resulting in undetectable HbA1c by the central laboratory, or hemolytic anemia requiring transfusion of blood or plasma products within 3 months before screening.
* Participants experienced with any severe hypoglycemic episode resulting in seizure, unconsciousness, or coma, and/or leading to hospitalization during the past 6 months before screening.
* Participants with insufficient smart phone skills or unwilling to properly use the virtual tools deemed by the investigator based on the observation and experiences over the digital screening procedure-Mental disorders or any neurologic disorder that would affect participant's ability to meet the study requirements, or participants deemed unlikely to safely manage insulin dosage by the investigator.
* Known hypersensitivity/intolerance to insulin glargine, rapid-acting insulin analogs or any of their excipients.
* Pregnant or breast-feeding women, or women who intend to become pregnant during the study period.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- United States (3):
  - Investigational Site Number 8400002, West Des Moines, Iowa
  - Investigational Site Number 8400004, Houston, Texas
  - Investigational Site Number 8400003, Bridgeport, West Virginia
- Canada (3):
  - Investigational Site Number 1240001, Barrie
  - Investigational Site Number 1240003, Oakville
  - Investigational Site Number 1240002, Thornhill

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 6 sites in Canada and United States between 19 September 2017 and 02 October 2018.
Pre-assignment Details: A total of 15 participants were randomized in study. Randomization was stratified by glycated hemoglobin (HbA1c) (less than [<] 7.6 percent [%] and greater than or equal to [>=] 7.6%) value at screening visit. Assignment in arms was done using interactive response technology (IRT) in 1:1 ratio to either virtual or traditional approach group.
Period: Overall Study
Arm/Group | Virtual | Traditional
Started (Randomized population) | 8 | 7
Safety Population (Treated) | 8 | 6
Completed | 5 | 4
Not Completed | 3 | 3
Not completed — Poor Compliance to Protocol | 0 | 2
Not completed — Study Terminated By Sponsor | 2 | 1
Not completed — Other than specified above | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population which included any participant who was allocated to a study conduct approach group regardless of whether the study conduct approach group was followed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual | Traditional | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (5.6) | 45.6 (14.3) | 49.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per meter square (kg/m^2)] — Population: Number analyzed signifies participants evaluable for this baseline measure.
  kilogram per meter square (kg/m^2)
    number analyzed (Participants) | 7 | 6 | 13
    (all) | 38.2 (18.4) | 30.9 (4.1) | 34.8 (13.8)
Duration of Type 1 Diabetes [Mean (Standard Deviation); unit: years] | 32.4 (11.5) | 19.3 (12.7) | 26.3 (13.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Hemoglobin A1c (HbA1c) to Week 24
Description: Change in HbA1c was calculated by subtracting baseline value from Week 24 value.
Time Frame: Baseline, Week 24
Population: Analysis was performed on intent to treat (ITT) population which included all randomized participants, irrespective of the trial approach group actually being used, analyzed according to the approach group allocated by randomization. Here, "overall number of participants analyzed" signifies participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 5 | 3
percentage of HbA1c | 0.10 (0.76) | 0.33 (0.57)

2. Secondary Outcome: Change From Baseline in Glycated Hemoglobin A1c to Week 16
Description: Change in HbA1c was calculated by subtracting baseline value from Week 16 value.
Time Frame: Baseline, Week 16
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' signifies participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 6 | 4
percentage of HbA1c | 0.23 (0.52) | 0.45 (0.13)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) to Week 16 and Week 24
Description: Change in FPG was calculated by subtracting baseline value from Week 16 value (for change at Week 16) and Week 24 (for change at Week 24) value.
Time Frame: Baseline, Week 16, Week 24
Population: Analysis was performed on ITT population. Here, "number analyzed" signifies participants with available data for each time point.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 8 | 7
millimole per liter (mmol/L)
  Week 16: number analyzed (Participants) | 5 | 4
  Week 16 | -0.660 (2.387) | -0.200 (4.555)
  Week 24: number analyzed (Participants) | 4 | 3
  Week 24 | -3.625 (3.406) | 2.900 (1.758)

4. Secondary Outcome: Participant Satisfaction With Trial Experience: Was It Worth It (WIWI) Questionnaire Response at Week 24
Description: Participant satisfaction with trial experience was measured using the WIWI questionnaire. The WIWI had 5 questions, 3 questions with level categorical response (Yes, No, and Unsure) scale, 1 question with 3 possible answers as: Better than I expected/The same as I expected/Worse than I expected, and 1 question with 3 possible answers: It improved/Stayed the same/Become worse.
Time Frame: At Week 24
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Work Productivity and Impairment-Study Participation (WPAI-SP) Scores to Week 24
Description: Effect of trial on a participants' ability to work and perform regular activities were measured using WPAI-SP. WPAI-SP had 6 items scored separately, where higher score indicated greater impairment and less productivity.
Time Frame: Baseline, Week 24
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Overall Study Experience-Participation (OSEP) Part-1 Questionnaire Score to Week 24
Description: Participant burden with trial participation was measured using the OSEP Questionnaire, administered electronically. OSEP Part-1 contained 4 items to examine perceptions of study participation. Each item was measured on an 11 point scale ranged from 0 (completely disagree) to 10 (completely agree), where higher score indicated higher perception of diabetes control.
Time Frame: Baseline, Week 24
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Overall Study Experience-Participation Part-2 Questionnaire Score to Week 24
Description: Participant burden with trial participation was measured using the OSEP Questionnaire, administered electronically. OSEP Part-2 contained 9 items to examine perceptions of study participation. Each item was measured on an 11 point scale ranged from 0 (completely disagree) to 10 (completely agree), where higher score indicated higher burden with trial participation.
Time Frame: Baseline, Week 24
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Resource Use Questionnaire (RUQ) Scores
Description: Healthcare resource use was measured using the RUQ which asked participants to report the resources used (time and expenses) during the previous 4 weeks in terms of visits to healthcare professionals.
Time Frame: During 24 weeks treatment period
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Diabetes Treatment Satisfaction Questionnaire Status (DTSQs) to Week 24
Description: The DTSQs was a validated questionnaire to assess participant's satisfaction with their diabetes treatment. It consisted of 8 items that were answered on a Likert scale from 0 (no satisfaction) to 6 (high satisfaction with treatment). Total treatment satisfaction score was the sum of items 1, 4-8 scores and ranged from 0 (no satisfaction) to 36 (high satisfaction with treatment).
Time Frame: Baseline, Week 24
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Diabetes Treatment Satisfaction Questionnaire Change (DTSQc) Score to Week 24
Description: DTSQc measured the relative change in treatment satisfaction from previous therapy. It consists of 8 items that were answered on a 6 point scale ranges from 3 (much less satisfied) to -3 (much more satisfied). Total treatment satisfaction score was the sum of items 1, 4-8 scores and ranged from -18 (much less satisfied) to +18 (much more satisfied), higher score indicated more satisfaction.
Time Frame: Baseline, Week 24
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Hypoglycemia Fear Survey-II (HFS-II) Scores
Description: Fear of hypoglycemia was measured with HFS-II at Week 24. The HFS-II comprises 33 items: 15 items explore behaviors that participants were engaged in to avoid low blood sugar and its negative consequences and 18 items related to concern/worry that participants had about their hypoglycemia. Responses to each item were made on a 5-point Likert scale ranges from 0 equal (=) "Never" to 4 = "Always". Total HFS mean score was determined by computing the mean of all 33 items and the score ranged from 0 to 4, where higher score indicated more fear/worry.
Time Frame: At Week 24
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Diabetes Distress Scale (DDS) Scores
Description: Diabetes-related distress was measured using DDS. The DDS contained 17 items related to potential problem areas that people with diabetes may experience. Participants were asked to consider the degree to which each of the items might have distressed or bothered them during the past month, and respond for each item on a 7 point scale ranges from 1 (not a problem) to 6 (a very serious problem), higher score indicated more diabetes related distress.
Time Frame: Week 0, Week 24
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in 7-Point Self-Monitoring of Plasma Glucose (SMPG) Profiles at Week 16 and Week 24 Per Time Point
Description: 7-point SMPG profiles were measured at the following 7 points at each visit (Baseline, Week 16, and Week 24): before breakfast, 2 hours after breakfast, before lunch, 2 hours after lunch, before dinner, 2 hours after dinner, and bedtime. For each time point, the value at each visit was calculated as the average of values obtained for the same time point across profiles performed in the week before the visit.
Time Frame: Baseline, Week 16, Week 24
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Average Daily Insulin Doses
Description: Average daily insulin doses included basal insulin doses, mealtime insulin doses, and total insulin doses.
Time Frame: During 24 weeks treatment period
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Overall Study Experience-Sites (OSES) Questionnaire Part-1: Hours Spent by Investigator
Description: An OSES questionnaire was completed by Site Investigator and had 2 parts. The OSES Part-1 contained quantitative 1 item (question) to examine resource requirements which was: Approximately how much time did you spend with this participant (in person or via phone) during this scheduled visit/communication? (hours)
Time Frame: During 24 weeks treatment period
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Overall Study Experience-Sites Questionnaire Part-2 Scores for Site-Perceived Participant Relationship and Satisfaction at Week 24
Description: An OSES questionnaire was completed by site investigator and had two parts. OSES Part-2 contains 2 items to examine investigator-participant relationship and satisfaction with care. Both items were assessed on a scale of 0 [completely disagree] to 10 [completely agree]), where highest score indicated a good relationship and satisfaction with care.
Time Frame: At Week 24
Population: Data were not collected due to data transfer issues therefore analysis was not performed for this outcome.
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Participants With At Least One Hypoglycemic Events (Any, Severe Documented Symptomatic, Probable Symptomatic, Asymptomatic, Pseudo-hypoglycemia: Any Time of the Day) During 24 Week Treatment Period
Description: Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Documented symptomatic hypoglycemia: an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <=3.9 mmol/L (70 mg/dL) or <3.0 mmol/L (54 mg/dL). Asymptomatic hypoglycemia: an event not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose concentration <=3.9 mmol/L (70 mg/dL) or <3.0 mmol/L (54 mg/dL). Probable symptomatic hypoglycemia: an event during which symptoms of hypoglycemia were not accompanied by plasma glucose determination but was presumably caused by a plasma glucose concentration. Pseudo-hypoglycemia: an event with any of the typical symptoms of hypoglycaemia with plasma glucose concentration >3.9 mmol/L (70 mg/dL).
Time Frame: During 24 weeks treatment period
Population: Analysis was done on safety population which included all randomized participants who did actually receive at least one dose of investigational medicinal product (IMP), regardless of the amount of IMP administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual | Traditional
Number analyzed (Participants) | 8 | 6
Participants
  Any hypoglycemia | 7 | 3
  Severe hypoglycemia | 0 | 0
  Documented symptomatic hypoglycemia: <=3.9 mmol/L | 6 | 3
  Documented symptomatic hypoglycemia: <3.0 mmol/L | 4 | 3
  Probable symptomatic hypoglycemia | 0 | 0
  Asymptomatic hypoglycemia <=3.9 mmol/L | 4 | 3
  Asymptomatic hypoglycemia <3.0 mmol/L | 1 | 1
  Pseudo-hypoglycemia >3.9 mmol/L | 1 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from time of first dose of study drug up to 25 weeks regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment emergent AEs that developed/worsened during the 'on treatment period' (from the first IMP administration to the last study drug administration + 1 week). Analysis was performed on safety population.
Arm/Group | Virtual | Traditional
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/6
Other Adverse Events (participants affected / at risk) | 2/8 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Virtual (N=8) | Traditional (N=6)
Obstructive Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Escherichia Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Virtual (N=8) | Traditional (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral Osteophyte (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intermittent Claudication (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Planned analysis could not be performed due to early study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT03260868/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03260868/SAP_001.pdf